CLINICAL TRIAL: NCT02788604
Title: Improving Quality of Life of Children With Cancer Through Psychosocial Screening and Improved Communication in Health Care Providers
Brief Title: Improving Quality of Life of Children With Cancer Through Psychosocial Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Provincial Health Services Authority British Columbia (Other)
Responsible Party: Principal Investigator, Maru Barrera, Psychologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 702843
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Cancer
Keywords: psychosocial screening, quality of life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants in this arm will have a summary of their family's psychosocial risk factors provided to the treatment team. This will occur twice: once shortly after diagnosis (within 2-4 weeks) and once approximately 6 months following diagnosis.
  Interventions: Other: Summary of psychosocial risk factors
- Control Group (Active Comparator): Participants in this arm will NOT have a summary of their family's psychosocial risk factors provided to the treatment team shortly after diagnosis. However, the risk factors will be distributed to the treatment team 6 months following diagnosis.
  Interventions: Other: Control

INTERVENTIONS:
Other: Summary of psychosocial risk factors — The treatment team will receive a psychosocial risk summary shortly following diagnosis based on parent report.
  Arms: Experimental Group
Other: Control — The treatment team will NOT receive a psychosocial risk summary shortly following diagnosis based on parent report.
  Arms: Control Group

SUMMARY:
In Canada, approximately 1450 children are diagnosed with cancer annually. Diagnosis of childhood cancer and its aggressive treatment can have devastating psychosocial effects on the whole family (e.g. unpleasant feelings or emotions that impact your daily activities). It is not known whether health care providers who treat these children use and value psychosocial tools or how beneficial the use of these tools is for these families. This research team will test the benefits of using psychosocial screening on the quality of life of treated children, parents and siblings.

DETAILED DESCRIPTION:
In Canada approximately 1450 children are diagnosed with cancer annually. Childhood cancer diagnosis and treatment can have devastating psychosocial effects on the family. Tools to screen for psychosocial risks (PSR) in pediatric oncology are rare. Our preliminary work adapted the Psychosocial Assessment Tool (PAT) for the Canadian population, PATrevised (PATrev), and developed the Psychosocial Care Checklist (PCCL). The PATrev is completed by parents of children with cancer, and yields a summary of the psychosocial needs of the patient, parents, and siblings. The PCCL assesses HCPs knowledge of family's psychosocial needs and services. Importantly, psychosocial screening is associated with reduced parental anxiety and improved child's quality of life (QOL). Demonstration of the tool's ability to maximize patient and family psychosocial outcomes is needed. Participants will be parents of children newly diagnosed with cancer, (patients and siblings (> 8 years), if available). Design: RCT with concealed allocation to experimental group (EG) and control group (CG), with repeated measures (after diagnosis= T1, 6 months later=T2). The EG treating team will receive a summary of PATrev risk information based on parent report. No risk information will be provided in the CG. Parents in both groups will complete the PATrev, family environment questionnaire, self--report and proxy reported QoL, distress and mood measures for the patient and one sibling. Patients and siblings will self-report on QOL, distress and mood. Patient charts will be reviewed (T2) to determine treatment intensity and documented psychosocial services for each family.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children newly diagnosed with cancer, within 2 to 4 weeks post-diagnosis.
* Siblings of children newly diagnosed with cancer, within 2-4 weeks post-diagnosis, between the ages of 8 years and 16 years, able to complete outcome measures, without a physical chronic condition.
* Children with cancer, newly diagnosed, within 2 to 4 weeks post-diagnosis, between the ages of 8 and 16 years, able to complete outcome measures.

Exclusion Criteria:

* Parents of children not diagnosed with cancer.
* Sibling of children not diagnosed with cancer
* Children not diagnosed with cancer.

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline psychological distress at pediatric cancer diagnosis to six months later | T1 (2-4 weeks following pediatric cancer diagnosis); T2 (6 months following diagnosis)
  Measured by Hospital Anxiety and Depression Scale (HADS). A standardized measure of symptoms of anxiety and depression in adults. The HADS is suitable for all ages from 17+. The HADS consists of 14 questions, which are ranked according to a 4 point Likert type scale.

SECONDARY OUTCOMES:
Change from baseline quality of life at pediatric cancer diagnosis to six months (Parent Self-Report) | T1 (2-4 weeks following pediatric cancer diagnosis); T2 (6 months following diagnosis)
  Measured by Caregiver Quality of Life Scale (CQOLC), 35 items using a five-point Likert-type scale to assess QoL in the family caregiver of cancer patients.
Change from baseline distress at pediatric cancer diagnosis to six months following | T1 (2-4 weeks following pediatric cancer diagnosis); T2 (6 months following diagnosis)
  Measured by the Distress Thermometer, a standardized screening tool for measuring emotional distress in adults. Has been widely used as a screening tool of distress in adult cancer patients and caregivers.
Change from baseline family climate at pediatric cancer diagnosis to six months | T1 (2-4 weeks following pediatric cancer diagnosis); T2 (6 months following diagnosis)
  Measured by Family Environment Scale (FES), a standardized measure of social climate within the family. The FES is a self-report measure which contains 27 true/false statements.
Change from baseline quality of life at pediatric cancer diagnosis to six months (Self) report | T1 (2-4 weeks following pediatric cancer diagnosis); T2 (6 months following diagnosis)
  Measured by Pediatric Quality of Life (PedsQL 4.0) - Cancer Module, Standardized tool measures child/parent perceptions of a child's health-related quality of life specific to having cancer. Self report and parent proxy perception of health-related quality of life across 8 domains: pain, nausea, procedure, and treatment anxiety, worry, cognition, physical and commutation.
Change from baseline quality of life at pediatric cancer diagnosis to six months (Proxy Report) | T1 (2-4 weeks following pediatric cancer diagnosis); T2 (6 months following diagnosis)
  Measured by Pediatric Quality of Life (PedsQL 4.0) - Generic Module.The measure assesses perception for the child's general health across global, physical, emotional , social and academic domains. Parent/self report by healthy sibling
Pediatric Distress Thermometer | T1 (2-4 weeks following pediatric cancer diagnosis); T2 (6 months following diagnosis)
  Standardized screening tool for measuring emotional distress in children. The distress thermometer adapted for pediatric population. Participants self-report on their distress on a line drawing representation of a thermometer. For this age group, distress is defined as worry, anxiety, sadness and fear on a visual analog scale from 0 (no distress) to 5 (moderate distress) to 10 (high distress). For patient with cancer and healthy sibling.
Pediatric Index of Emotional Distress (PI-ed) | T1 (2-4 weeks following pediatric cancer diagnosis); T2 (6 months following diagnosis)
  A 14-item self-report measure of emotional distress in children rated on a 4-point Likert scale (0 = not at all; 3 = always). This measure, based on the Hospital Anxiety and Depression Scale (HADS;[62]), was designed to differentiate symptoms of emotional distress from physical illness in pediatric populations. It comprises two subscales assessing depression and anxiety, which when summated, provides a global index of emotional distress. For child with Cancer and healthy sibling.

CONTACTS AND LOCATIONS:
Overall Officials: Maru Barrera, PhD, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Canada (2):
  - BC Women and Children's Hospital, Vancouver, British Columbia
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boman K, Lindahl A, Bjork O. Disease-related distress in parents of children with cancer at various stages after the time of diagnosis. Acta Oncol. 2003;42(2):137-46. doi: 10.1080/02841860310004995. PMID 12801132
- [Background] Kazak AE, Simms S, Rourke MT. Family systems practice in pediatric psychology. J Pediatr Psychol. 2002 Mar;27(2):133-43. doi: 10.1093/jpepsy/27.2.133. PMID 11821497
- [Background] Sawyer MG, Antoniou G, Toogood I, Rice M, Baghurst PA. A prospective study of the psychological adjustment of parents and families of children with cancer. J Paediatr Child Health. 1993 Oct;29(5):352-6. doi: 10.1111/j.1440-1754.1993.tb00533.x. PMID 8240863
- [Background] Wijnberg-Williams BJ, Kamps WA, Klip EC, Hoekstra-Weebers JE. Psychological distress and the impact of social support on fathers and mothers of pediatric cancer patients: long-term prospective results. J Pediatr Psychol. 2006 Sep;31(8):785-92. doi: 10.1093/jpepsy/jsj087. Epub 2005 Oct 26. PMID 16251479
- [Background] Woodgate RL, Degner LF, Yanofsky R. A different perspective to approaching cancer symptoms in children. J Pain Symptom Manage. 2003 Sep;26(3):800-17. doi: 10.1016/s0885-3924(03)00285-9. PMID 12967729
- [Background] Kupst MJ, Natta MB, Richardson CC, Schulman JL, Lavigne JV, Das L. Family coping with pediatric leukemia: ten years after treatment. J Pediatr Psychol. 1995 Oct;20(5):601-17. doi: 10.1093/jpepsy/20.5.601. PMID 7500233
- [Background] Barrera M, D'Agostino NM, Gibson J, Gilbert T, Weksberg R, Malkin D. Predictors and mediators of psychological adjustment in mothers of children newly diagnosed with cancer. Psychooncology. 2004 Sep;13(9):630-41. doi: 10.1002/pon.765. PMID 15334531
- [Background] Kazak AE, Brier M, Alderfer MA, Reilly A, Fooks Parker S, Rogerwick S, Ditaranto S, Barakat LP. Screening for psychosocial risk in pediatric cancer. Pediatr Blood Cancer. 2012 Nov;59(5):822-7. doi: 10.1002/pbc.24166. Epub 2012 Apr 10. PMID 22492662
- [Background] Barrera M, Hancock K, Rokeach A, Cataudella D, Atenafu E, Johnston D, Punnett A, Nathan PC, Bartels U, Silva M, Cassidy M, Jansen P, Shama W, Greenberg C. External validity and reliability of the Psychosocial Assessment Tool (PAT) among Canadian parents of children newly diagnosed with cancer. Pediatr Blood Cancer. 2014 Jan;61(1):165-70. doi: 10.1002/pbc.24774. Epub 2013 Sep 17. PMID 24106172
- [Background] Patel SK, Mullins W, Turk A, Dekel N, Kinjo C, Sato JK. Distress screening, rater agreement, and services in pediatric oncology. Psychooncology. 2011 Dec;20(12):1324-33. doi: 10.1002/pon.1859. Epub 2010 Oct 5. PMID 20925136
- [Derived] Barrera M, Young MA, Hancock K, Chung J. Early trajectory of psychosocial risk in families of children and adolescents newly diagnosed with cancer. Support Care Cancer. 2022 Feb;30(2):1815-1822. doi: 10.1007/s00520-021-06581-3. Epub 2021 Oct 4. PMID 34608532
- [Derived] Barrera M, Alexander S, Atenafu EG, Chung J, Hancock K, Solomon A, Desjardins L, Shama W, Mills D. Psychosocial screening and mental health in pediatric cancer: A randomized controlled trial. Health Psychol. 2020 May;39(5):381-390. doi: 10.1037/hea0000825. Epub 2020 Jan 23. PMID 31971403
- [Derived] Barrera M, Hancock K, Atenafu E, Alexander S, Solomon A, Desjardins L, Shama W, Chung J, Mills D. Quality of life in pediatric oncology patients, caregivers and siblings after psychosocial screening: a randomized controlled trial. Support Care Cancer. 2020 Aug;28(8):3659-3668. doi: 10.1007/s00520-019-05160-x. Epub 2019 Dec 6. PMID 31811485